CLINICAL TRIAL: NCT01991275
Title: The Efficacy of Intrathecal Morphine in Patients Undergoing Robot-assisted Prostatectomy
Brief Title: Intrathecal Morphine in Robot-assisted Prostatectomy
Acronym: RoboITMProst
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Deok Man Hong, Associate professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ITMRoboProstDMHong
Record Dates: First submitted 2013-11-18; First posted 2013-11-25 (Estimated); Last update posted 2015-07-03 (Estimated); Status verified 2015-07

CONDITIONS: Prostatic Neoplasms
Keywords: Prostatic Neoplasms; Laparoscopy; Injections, Spinal; Morphine
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- The ITM group (Experimental): The postoperative pain management includes both the intrathecal morphine injection and the intravenous patient-controlled analgesia.
  Interventions: Drug: The intravenous patient-controlled analgesia; Drug: The intrathecal morphine injection
- The IV-PCA group (Placebo Comparator): The postoperative pain management includes only the intravenous patient-controlled analgesia.
  Interventions: Drug: The intravenous patient-controlled analgesia

INTERVENTIONS:
Drug: The intravenous patient-controlled analgesia — The intravenous injection of morphine using the patient-controlled analgesia machine
Drug: The intrathecal morphine injection — A single injection of morphine intrathecally
  Arms: The ITM group

SUMMARY:
This study will investigate the efficacy and safety of intrathecal morphine for the patients undergoing robot-assisted prostatectomy

DETAILED DESCRIPTION:
Prostatectomy is the treatment of choice for prostate cancer. The robot-assisted prostatectomy is becoming the most popular surgical method for prostate cancer. The small incision after robot-assisted prostatectomy is thought to reduce the postoperative pain. There is few investigations for the strategy to reduce the postoperative pain of robot-assisted prostatectomy.

The intrathecal morphine injection is known to reduce postoperative pain for surgeries like hepatectomy, myomectomy and open prostatectomy. This method, however, is not yet studied for the robot-assisted prostatectomy. This study will investigate the efficacy and safety of intrathecal morphine for the patients undergoing robot-assisted prostatectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for the open nephrectomy

Exclusion Criteria:

* Patients with renal insufficiency
* Patients with coagulopathy
* History of any neurologic disorder
* History of recent infection in 2 weeks
* History of drug abuse
* Patients who cannot understand the usage of th intravenous patient-controlled analgesia
* Patients using opioids due to the chronic pain

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-11; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
The evaluation of pain at 24 hours after surgery | at postoperatively 24 hours
  The doctor blinded to the investigation will visit patients. The pain will be assessed at rest and at coughing using visual analogue scale.

SECONDARY OUTCOMES:
The consumption of analgesics | at postoperatively 24 hours
  The total amount of opioids (IV morphine) used for 24 hours after surgery will be recorded and compared.
The consumption of intraoperative opioids | From the induction of anesthesia till the emergence of anesthesia, an expected average of 4 hours
  The total amount of intraoperative opioids (IV remifentanil) will be recorded and compared.
The side effects of opioids after surgery | During 72 hours after the end of surgery
  Any side effects of opioids including nausea, vomiting, dizziness, sedation, headache, pruritus and respiratory depression will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Deok-Man Hong, PhD, Study Director — Seoul National University of Hospital
Locations (1):
- Seoul National University of Hospital, Seoul, South Korea